CLINICAL TRIAL: NCT01566175
Title: Use of the Neovasc Coronary Sinus Reducer System for the Treatment of Refractory Angina Pectoris in Patients With Angina Class 3-4 Who Are Not Candidates for Revascularization
Brief Title: Use of the Neovasc Coronary Sinus Reducer System for the Treatment of Refractory Angina Pectoris in Patients With Ngina Class 3-4 Who Are Not Candidates for Revascularization
Acronym: Reducer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Shockwave Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Eli Sprecher, MD, Prof. Gad Keren, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neovasc Reducer
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Refractory Angina
Keywords: Neovasc Reducer; Coronary Sinus; Refractory Angina Pectoris; angina class 3-4
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neovasc coronary sinus reducer (Experimental): open label: Neovasc coronary sinus reducer
  Interventions: Device: Neovac coronary sinus reducer

INTERVENTIONS:
Device: Neovac coronary sinus reducer — reducer
  Other Names: Reducer

SUMMARY:
The purpose of this study is to implant the Reducer in patients with the symptoms of refractory angina, that suffer from refractory angina who demonstrate reversible ischemia.

DETAILED DESCRIPTION:
* Interventional, Allocation: Open label, Primary Purpose: Treatment
* Diagnosis and treatment for which the device is required:Patients with advanced obstructive coronary artery disease and severe disabling refractory angina despite optimal medical therapy. No revascularization option available.
* Why this unlicensed device is chosen over a licensed device or conventional therapies for this particular patient? Patient currently treated with optimal medical therapies that include: long acting nitrates, beta blockers, and calcium channel blockers. The patient is not amendable to re-do bypass graft surgery, not amendable to percutaneous coronary intervention, as determined by recent coronary angiography.

There is no other licensed device that can effectively ameliorate refractory angina and reduce the number of angina episodes and improve quality of life.

-The current device has been used in 25 patients to date. Safety information at 6 months had been published (JACC 2007;49:1783). Extended safety and efficacy information at 3 years had been reported in March 2010 (ACC Annual Scientific conference). The device has not been associated with any procedure-related adverse events during the follow-up period.

Risks (theoretical):•Coronary sinus dissection at the time of implantation. •Coronary sinus perforation and acute cardiac tamponade requiring drainage. •Device migration and embolization. •Late coronary sinus occlusion These risk were not reported in patients who receieved the device. Benefits: •Reduce angina severity. •Improve quality of life. •Reduction in the intensity of medical therapy with decrease side effects. •Reduced incidence of hospital admissions, emergency room visits and outpatient clinic visits for refractory angina. •Improved left ventricular function, and reduced LV end diastolic pressure. These patients have poor quality of life. They are disable and unable to work or to perform basic daily activities. Cannulation of the coronary sinus presents procedural risks similar to that of pacemaker electrode insertion, a procedure which is frequently performed in Interventional cardiology. For these particular patients with poor quality of life, the offered technology can potentially make them more active, more productive, and less dependent on medication and the health system.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Symptomatic CAD with chronic refractory angina pectoris classified as Canadian Cardiovascular Society (CCS) grade III or IV despite attempted optimal medical therapy for thirty days prior to screening
* Non-candidate for surgical or percutaneous coronary intervention, as determined by 2 independent Professors of Internal medicine
* Reversible ischemia of the left ventricular wall demonstrated by Dobutamine Stress Echocardiography (Dobutamine ECHO; DSE), or by Thallium Spect

Exclusion Criteria:

* Recent (within three months) acute coronary syndrome
* Recent (within six months) PCI or CABG
* Unstable angina (recent onset angina, crescendo angina, or rest angina with ECG changes) during the thirty days prior to screening
* De-compensated congestive heart failure or hospitalization due to CHF during the three months prior to screening
* Life threatening rhythm disorders or any rhythm disorders that would require placement of an internal defibrillator and or pacemaker
* Severe chronic obstructive pulmonary disease as indicated by a forced expiratory volume in one second that is less than 55% of the predicted value
* Severe valvular heart disease
* Patient with pacemaker or defibrillator electrode in the right atrium, right ventricle, or coronary sinus
* Patient having undergone tricuspid valve replacement or repair
* Known allergy to stainless steel or nickel
* Patient with anomalous or abnormal CS as demonstrated by angiogram. Abnormality defined as: Abnormal CS anatomy (e.g., tortuosity, aberrant branch, persistent left SVC) and/or; CS diameter at the site of implantation> 12mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-08-30 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Canadian Cardiovascular Society Angina Score | 6 months
  A decrease of two or more Canadian Cardiovascular Society Angina Score grades from baseline to six-month post-procedural evaluation in Reducer and Control groups

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Tel Aviv Medical Center, Tel Aviv